CLINICAL TRIAL: NCT01302587
Title: A Prospective, Open Label, Assessment of [an Albuterol] Hydrofluoroalkane (HFA) Metered Dose Inhaler MDI Integrated Dose Counter
Brief Title: A Study to Evaluate the Integrated Dose Counter on an Albuterol Hydrofluoroalkane (HFA) Metered Dose Inhaler (MDI)
Status: Completed | Type: Observational
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ABM-AS-307
Record Dates: First submitted 2011-02-16; First posted 2011-02-24 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD); Emphysema; Chronic Bronchitis
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic | interventions — Albuterol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Albuterol MDI: All participants in this study will receive an albuterol MDI inhaler.
  Interventions: Drug: Albuterol

INTERVENTIONS:
Drug: Albuterol — Albuterol MDI with integrated dose counter. Each participant will use 2 oral inhalations of 90 micrograms each of albuterol twice a day for the length of the study.

SUMMARY:
This study is evaluating the effectiveness of a dose counter for an inhaler device used to deliver medication to people diagnosed with asthma or COPD.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent
* General good health
* Asthma or COPD
* Capable of understanding the requirements, risks, and benefits of study participation.
* Able to demonstrate proper metered-dose inhaler use and technique.
* Other inclusion criteria apply

Exclusion Criteria:

* History of life-threatening asthma or COPD that is defined for this protocol as an asthma or COPD episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures.
* Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 2 weeks of Screening Visit.
* Is being treated with a long-acting β2-agonist alone.
* Is currently being treated with Ventolin HFA.
* Any asthma or COPD exacerbation requiring oral corticosteroids within 2 months of Screening Visit. A subject must not have had any hospitalization for asthma or COPD within 4 months prior to Screening Visit.
* Historical or current evidence of a clinically significant non-asthmatic acute or chronic condition.
* Uncontrolled hypertension
* History of any adverse reaction to any component of the HFA-MDI formulation.
* Participation in any investigational drug study within the 30 days preceding the Screening Visit.
* Other exclusion criteria apply.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People diagnosed with asthma or Chronic Obstructive Pulmonary Disease (also known as COPD, emphysema or chronic bronchitis)
Sampling Method: Non-Probability Sample
Enrollment: 306 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The number of times the counter advanced but the inhaler did not actuate | Days 1 through 46
  MDI actuates but the counter display does not advance.

SECONDARY OUTCOMES:
The number of times the inhaler actuated but the counter did not advance. | Days 1 through 46
  Counter advances but the MDI does not actuate.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Leader, Study Director — Teva Respiratory R&D
Locations (25):
- United States (25):
  - Teva Clinical Study Site, Glendale, Arizona
  - Teva Clinical Study Site 10100, Mission Viejo, California
  - Teva Clinical Study Site 10093, Orange, California
  - Teva Clinical Study Site 10089, San Diego, California
  - Teva Clinical Study Site 10098, Wheat Ridge, Colorado
  - Teva Clinical Study Site, Miami, Florida
  - Teva Clinical Study Site 10082, Ormond Beach, Florida
  - Teva Clinical Study Site, Tamarac, Florida
  - Teva Clinical Study Site 10090, Indianapolis, Indiana
  - Teva Clinical Study Site 10097, Overland Park, Kansas
  - Teva Clinical Study Site 10087, Wichita, Kansas
  - Teva Clinical Study Site, Fall River, Massachusetts
  - Teva Clinical Study Site 10094, North Dartmouth, Massachusetts
  - Teva Clinical Study Site 10086, Minneapolis, Minnesota
  - Teva Clinical Study Site 10083, High Point, North Carolina
  - Teva Clinical Study Site 10092, Raleigh, North Carolina
  - Teva Clinical Study Site 10085, Canton, Ohio
  - Teva Clinical Study Site 10080, Tulsa, Oklahoma
  - Teva Clinical Study Site 10088, Eugene, Oregon
  - Teva Clinical Study Site 10095, Portland, Oregon
  - Teva Clinical Study Site 10081, Greenville, South Carolina
  - Teva Clinical Study Site 10084, Spartanburg, South Carolina
  - Teva Clinical Study Site, Dallas, Texas
  - Teva Clinical Study Site 10091, New Braunfels, Texas
  - Teva Clinical Study Site 10099, Seattle, Washington

REFERENCES:
- [Derived] Given J, Taveras H, Iverson H, Lepore M. Prospective, open-label assessment of albuterol sulfate hydrofluoroalkane metered-dose inhaler with new integrated dose counter. Allergy Asthma Proc. 2013 Jan-Feb;34(1):42-51. doi: 10.2500/aap.2012.33.3647. Epub 2012 Dec 20. PMID 23265285